CLINICAL TRIAL: NCT06255639
Title: Biomechanical and Metabolic Assessment Pre and Post Vertebroplasty in Multiple Myeloma Patients With Vertebral Collapse
Status: Recruiting | Type: Observational
Sponsor: Centro di Riferimento Oncologico - Aviano (Other)
Responsible Party: Sponsor
Other Study IDs: CRO-2020-35
Record Dates: First submitted 2024-01-19; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MM patient candidate to vertebroplasty

SUMMARY:
In patients with Multiple Myeloma (MM), bone lesions can lead to multiple vertebral lesions, with vertebral collapses. The introduction of minimally invasive procedures such as percutaneous vertebroplasty allow patients to return to a fair level of function and a significant reduction in pain. Despite medical therapies, radiotherapy, analgesics and vertebroplasty procedures, patients with multiple spinal injuries often complain of pain and stiffness that limit their mobility, daily activities and work. The aim of this study is to measure how the biomechanical, thermo-metabolic and algic parameters change after vertebroplasty in patients with MM

DETAILED DESCRIPTION:
In patients with Multiple Myeloma (MM), bone lesions can lead to multiple vertebral lesions, with vertebral collapses. The introduction of minimally invasive procedures such as percutaneous vertebroplasty allow patients to return to a fair level of function and a significant reduction in pain. Despite medical therapies, radiotherapy, analgesics and vertebroplasty procedures, patients with multiple spinal injuries often complain of pain and stiffness that limit their mobility, daily activities and work. The aim of this study is to measure how the biomechanical, thermo-metabolic and algic parameters change after vertebroplasty in patients with MM

ELIGIBILITY:
Inclusion Criteria:

* Age≥ 18 years;
* Diagnosis of multiple myeloma;
* Clinical indication and eligibility for vertebroplasty procedure;
* Performance Status (ECOG) 0-2;
* Life expectancy greater than three months;
* Low-resolution full skeletal CT scan at disease onset and/or at follow-up;
* Spine pain with stiffness and functional impediment pre vertebroplasty;
* Able to express appropriate consent for participation in the study (e.g. Able to understand Italian, patient with intact cognitive abilities)

Exclusion Criteria:

* presence of spinal cord compressions;
* unstable spinal injuries, requiring an orthopaedic back brace;
* risk of spinal cord injury;
* body mass index BMI>28 kg/m2.
* absence of signed informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from multiple myeloma (MM) with multiple vertebral lesions and candidates for vertebroplasty, consecutively diagnosed with MM in the period from 2015 to 2021 at the study center
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-10-15 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Difference in mean of kinematic data for walking before and after vertebroplasty | 2 months
  Difference in mean of kinematic data for walking before and after vertebroplasty
difference in mean of movement range for affected joints before and after vertebroplasty | 2 months
  difference in mean of movement range for affected joints before and after vertebroplasty
Difference in mean of energy expenditure before and after vertebroplasty | 2 months
  Difference in mean of energy expenditure before and after vertebroplasty

SECONDARY OUTCOMES:
To explore the impact of vertebroplasty on thermal parameters | 2 months
  Central and superficial temperature will be measured before and after vertebroplasty. Difference will be reported as intrapatient mean difference
To explore the impact of vertebroplasty on metabolic parameters | 2 months
  Carbon dioxide production after 30 minutes of walking will be measured before and after vertebroplasty and intrapatient mean difference will be reported.
To explore the impact of vertebroplasty on metabolic parameters | 2 months
  Cardiac frequency after 30 minutes of walking will be measured before and after vertebroplasty and intrapatient mean difference will be reported.
To explore the impact of vertebroplasty on metabolic parameters | 2 months
  Oxygen consumption after 30 minutes of walking will be measured before and after vertebroplasty and intrapatient mean difference will be reported.
To explore the impact of vertebroplasty on pain | 2 months
  Perceived pain will be measured using the Brief Pain Inventory scale (BPI) before and after vertebroplasty. Difference will be reported as intrapatient mean difference. BPI values range between 0 and 10, with higher scores meaning worst pain

CONTACTS AND LOCATIONS:
Overall Officials: Mariagrazia Michieli, MD, Principal Investigator — Centro di Riferimento Oncologico (CRO) di Aviano - IRCCS
Locations (1):
- Centro di Riferimento Oncologico (CRO) di Aviano - IRCCS, Aviano, Pordenone, Italy